CLINICAL TRIAL: NCT02824458
Title: A Multicenter, Randomized,Double-Blind Study of Gefitinib in Combination With Apatinib or Placebo in Previously Untreated Patients With EGFR Mutation-Positive Advanced Non-squamous Non-Small-Cell Lung Cancer
Brief Title: A Study of Gefitinib With or Without Apatinib in Patients With Advanced Non-squamous Non-Small-Cell Lung Cancer Harboring EGFR Mutations
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hongyun Zhao, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-FXY-023
Record Dates: First submitted 2016-06-23; First posted 2016-07-06 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: EGFR Tyrosine Kinase Inhibitors Plus VEGFR Inhibitors
Keywords: EGFR tyrosine kinase inhibitors; VEGFR inhibitor; NSCLC
MeSH Terms: interventions — apatinib; Gefitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gefitinib + Apatinib (Experimental): (Part A) Phase I, Open-label, Dose-escalation Study Escalating doses(500mg, 750mg, or 250mg) of Apatinib in combination with 250mg Gefitinib daily orally. Participants may continue to receive treatment until progress or intolerable.
  (Part B)Multicenter, Randomized, Double-Blind Study Apatinib (dose determined from Part A of study) in combination with 250mg Gefitinib.
  Interventions: Drug: Apatinib; Drug: Gefitinib
- Gefitinib + Placebo (Placebo Comparator): (Part A) Not Applicable
  (Part B) Placebo in combination with 250mg Gefitinib. Participants may continue to receive treatment until progress or intolerable.
  Interventions: Drug: Gefitinib; Drug: Placebo

INTERVENTIONS:
Drug: Apatinib — Patients will be treated with Apatinib, 250/500/750 mg(dose determined from Part A of study) p.o., daily
  Other Names: YN968D1
  Arms: Gefitinib + Apatinib
Drug: Gefitinib — Patients will be treated with Gefitinib, 250 mg p.o., daily
  Other Names: Iressa
Drug: Placebo
  Arms: Gefitinib + Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of Apatinib in combination with Gefitinib as compared to placebo in combination with Gefitinib in participants with stage ⅢB-IV Non-squamous non-small-cell lung cancer (NSCLC) harboring an activating epidermal growth factor receptor (EGFR) mutation (Del19 and L858R). Safety and tolerability of Apatinib in combination with Gefitinib will be assessed in the first portion (Part A) before proceeding to the second portion of this study (Part B).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 and ≤ 70 years of age
2. Eastern Cooperative Oncology Group(ECOG)performance scale 0 - 1.
3. Life expectancy of more than 3 weeks.
4. Histologically or cytologic confirmed，locally advanced and/or metastatic non-squamous NSCLC of stage IIIB (unsuitable for radiotherapy) or IV or recurrent NSCLC; At least one measurable lesion according to RECIST 1.1 which has not received radiotherapy or cryotherapy.
5. Documented evidence of tumor harboring an activating EGFR mutation (Example 19 del and L858R) .
6. None previous chemotherapy or targeted therapy. NOTE: neoadjuvant and/or adjuvant therapy is allowed which is completed before 6 months.
7. Prior radiation therapy is allowed if: 25% or less of total bone marrow had been irradiated,pelvis and chest had not been irradiated; at least 4 weeks have elapsed from the completion of radiation treatment, and the acute toxicity from radiation treatment had been recover; irradiated lesion is not including measurable lesions unless documented progress after radiation.
8. Adequate hepatic, renal, heart, and hematologic functions (Absolute Neutrophil Count(ANC) ≥ 1.5×109/L, Platelet (PLT) ≥ 100×109/L, Hemoglobin(HB) ≥ 100 g/L, total bilirubin within 1.5×the upper limit of normal(ULN), and serum transaminase≤2.5×the Upper Limit Of Normal(ULN), serum creatine ≤ 1 x Upper Limit Of Normal(ULN), creatinine clearance rate ≥ 50ml/min,
9. For women of child-bearing age, the pregnancy test results (serum or urine) within 7 days before enrolment must be negative. They will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men (previous surgical sterilization accepted), will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug.
10. Signed and dated informed consent. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

1. Squamous cell carcinoma (including adenosquamous carcinoma, undifferentiated carcinoma); small cell lung cancer (including small cell and non-small cell mixed lung cancer)
2. Symptomatic brain metastases (Patients who have no symptoms and is not needed to receive therapy before 21 days may participate in this trial, but need to be confirmed by MRI\CT or venography that no hematencephalon symptom);
3. Radiologically documented evidence of major blood vessel invasion or encasement by cancer; Obvious cavity or necrosis formed in the tumor.
4. Uncontrolled hypertension(systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mm Hg) even though two or more than two hypotensive agents application.
5. Patients who suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female ≥ 470 ms). Grade III-IV cardiac insufficiency according to New York Heart Association(NYHA) criteria or echocardiography check: left ventricular ejection fraction (LVEF)<50%;
6. History of pulmonary interstitial diseases or concurrent pulmonary interstitial diseases.
7. Coagulation disfunction（INR>1.5 o rPT>Upper Limit Of Normal(ULN)+4s or Activated Partial Thromboplastin Time (APTT) >1.5 Upper Limit Of Normal(ULN)）, hemorrhagic tendency or receiving the therapy of thrombolysis or anticoagulation.
8. History of clinically significant haemoptysis =< 2 months (more than 2.5ml or half of one tea spoon of fresh blood per day) prior to registration.
9. History of clinically relevant major bleeding event (e.g. gastrointestinal hemorrhage, bleeding gastric ulcer, occult blood test ≥ (++), and vasculitis ;
10. Within 6 months before the first treatment occurs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack(TIA), hematencephalon, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.
11. Known inherited and acquired hemorrhagic and thromboplastic possibility (such as hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc.)
12. Long-term untreated wounds or fractures.
13. Within 4 weeks of major surgery and/or injures, fractures , ulceration.
14. Significant factors that influence the ingestion and absorption of medicine, (e.g. unable swallow, chronic diarrhea and intestinal obstruction);
15. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess ≤ 6 months.
16. Urine protein≥++, or 24h urine protein quantitation≥1.0g;
17. Symptomatic serous effusion requiring treatment .(including hydrothorax, ascites, hydropericardium);
18. Active infection need antimicrobial treatments;
19. History of psychiatric drugs abuse and not be abstinent, or dysphrenia;
20. Less than 4 weeks from the last clinical trial
21. History or concomitant other malignancy except cured basal cell skin cancer, or carcinoma in situ of the cervix, or superficial bladder cancer;
22. Administration of strong/potent cytochrome P450 (CYP)3A4 inhibitors within 7 days, or inducers within 12 days;
23. Pregnant or breastfeeding women;
24. Other conditions regimented at investigators' discretion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2016-06; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
(Part A) Determine Dose-Limiting Toxicity (DLT) of Apatinib in combination with Gefitinib | 1 months
  Determine the safety, tolerability and DLTs of Apatinib in Combination With Gefitinib
(Part A) Maximum Tolerated Dose (MTD) of Apatinib in Combination With Gefitinib | 1 months
  MTD was determined by testing increasing doses up to 750 mg daily (qd) on dose escalation cohorts 1 to 3 with 3 patients each. MTD reflects highest dose of drug that did not cause an unacceptable side effect (= Dose Limiting Toxicity (DLT) in more than 30% of patients; e.g., hematologic toxicities like Common Toxicity Criteria (CTC) Grade 4 Neutropenia in specific conditions, platelets < 25,000 cells/mL; specific non-hematologic/biochemical toxicities CTC Grade 3 or 4; additionally, any toxicity considered by the investigator severe enough was designated a DLT); CTC Version 2 were used.
(Part B) Progression Free Survival (PFS) | Randomization to Measured Progressive Disease or Death from Any Cause (Estimated as 42 Months)
  Time from the date of enrolment until documented progression or death, whichever occurs first.

SECONDARY OUTCOMES:
(Part B) Overall Survival (OS) | Randomization to Date of Death from Any Cause (Estimated as 50 Months)
  Time from the date of enrolment until death from any cause.
(Part B) Objective Response Rate (ORR) | Randomization to Disease Progression (Estimated as 42 Months)
  Best overall response (complete remission or partial remission) across all assessment time-points according to RECIST Criteria 1.1, during the period from enrolment to termination of trial treatment
(Part B) Disease Control Rate (DCR) | Randomization to Disease Progression (Estimated as 42 Months)
  Achievement of objective response or stable disease for at least 6 weeks
(Part B) Duration of Response (DoR) | Date of Complete Response (CR) or Partial Response (PR) to Date of Objective Disease Progression or Death Due to Any Cause (Estimated as 42 Months)
  Interval from the date of first documentation of objective response by RECIST to the date of first documented progression or relapse
(Part B) Time to progression disease (TTPD) | Randomization to Measured Progressive Disease (Estimated as 42 Months)
  Time to progression disease
(Part B) Quality of Life (QoL) questionnaire | Baseline, End of Study (Estimated as 50 Months)
(Part A + B) Safety assessment : Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Randomization to Measured Progressive Disease (Estimated as 50 Months)
  including adverse events, physical examination, vital signs (including Blood Pressure(BP)), clinical chemistry and hematology
(Part A) Area Under roc Curve (last) | Apatinib & Gefitinib: Cycle1 Day 1 and 15
  Area under the plasma concentration time profile from time zero to the time of the last quantifiable concentration
(Part A) Area Under roc Curve (tau) | Apatinib & Gefitinib: Cycle1 Day 1 and 15
  Area under the plasma concentration time profile after single dose from time zero to the next dose
(Part A) Cmax | Apatinib & Gefitinib: Cycle1 Day 1 and 15
  Maximum observed plasma concentration
(Part A) Tmax | Apatinib & Gefitinib: Cycle1 Day 1 and 15
  Time for Cmax
(Part A) t½a | Apatinib & Gefitinib: Cycle1 Day 1 and 15
  Terminal half life
(Part A) Ctrough | Apatinib & Gefitinib: Cycle1 Day 1 and 15
  Predose concentration during multiple dosing
(Part A) The Apparent Clearance(CL/F) | Apatinib & Gefitinib: Cycle1 Day 1 and 15
  Apparent clearance
(Part A) The Apparent Volume of Distribution (Vd/F) | Apatinib & Gefitinib: Cycle1 Day 1 and 15
  Apparent volume of distribution
(Part A) The Metabolite to Parent Ratio of Area Under roc Curve (tau) | Apatinib & Gefitinib: Cycle1 Day 1 and 15
  Metabolite to parent ratio for Area Under roc Curve (tau)
(Part A) The Metabolite to Parent Ratio of Css,max(MRCmax) | Apatinib & Gefitinib: Cycle1 Day 1 and 15
  Metabolite to parent ratio for Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Hongyun Zhao, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao H, Yao W, Min X, Gu K, Yu G, Zhang Z, Cui J, Miao L, Zhang L, Yuan X, Fang Y, Fu X, Hu C, Zhu X, Fan Y, Yu Q, Wu G, Jiang O, Du X, Liu J, Gu W, Hou Z, Wang Q, Zheng R, Zhou X, Zhang L. Apatinib Plus Gefitinib as First-Line Treatment in Advanced EGFR-Mutant NSCLC: The Phase III ACTIVE Study (CTONG1706). J Thorac Oncol. 2021 Sep;16(9):1533-1546. doi: 10.1016/j.jtho.2021.05.006. Epub 2021 May 24. PMID 34033974
- [Derived] Deng Z, Qin Y, Liu Y, Zhang Y, Lu Y. Role of Antiangiogenic Agents Combined With EGFR Tyrosine Kinase Inhibitors in Treatment-naive Lung Cancer: A Meta-Analysis. Clin Lung Cancer. 2021 Jan;22(1):e70-e83. doi: 10.1016/j.cllc.2020.08.005. Epub 2020 Sep 18. PMID 33067126
- [Derived] Zhang Z, Zhang Y, Luo F, Ma Y, Fang W, Zhan J, Li S, Yang Y, Zhao Y, Hong S, Zhou T, Zhang Y, Zhao S, Huang Y, Zhao H, Zhang L. Dual blockade of EGFR and VEGFR pathways: Results from a pilot study evaluating apatinib plus gefitinib as a first-line treatment for advanced EGFR-mutant non-small cell lung cancer. Clin Transl Med. 2020 Jun;10(2):e33. doi: 10.1002/ctm2.33. Epub 2020 Jun 4. PMID 32508029
- [Derived] Zhang Z, Luo F, Zhang Y, Ma Y, Hong S, Yang Y, Fang W, Huang Y, Zhang L, Zhao H. The ACTIVE study protocol: apatinib or placebo plus gefitinib as first-line treatment for patients with EGFR-mutant advanced non-small cell lung cancer (CTONG1706). Cancer Commun (Lond). 2019 Nov 7;39(1):69. doi: 10.1186/s40880-019-0414-4. PMID 31699150